CLINICAL TRIAL: NCT05268289
Title: An Adaptive, Randomized, Double-blind, Dose Exploration, Parallel Group, Placebo Controlled, Multicenter Phase 2 Trial to Evaluate the Efficacy, Safety and Tolerability of LNP023 in Combination With Standard-of-care With and Without Oral Corticosteroids in Patients With Active Lupus Nephritis Class III-IV, +/- V
Brief Title: Study of Efficacy and Safety of LNP023 in Participants With Active Lupus Nephritis Class III-IV, +/- V
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNP023K12201; 2021-002046-33 (EudraCT Number)
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lupus Nephritis
Keywords: LNP023; Iptacopan; Lupus Nephritis; proteinuria; Urine Protein-to-Creatinine Ratio; complete renal response; estimated glomerular filtration rate; renal flares; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Nephritis; Proteinuria; Lupus Erythematosus, Systemic | interventions — iptacopan; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Iptacopan + standard of care (part 1) (Active Comparator): Iptacopan + standard of care
  Interventions: Drug: Iptacopan (part 1)
- Placebo matching iptacopan + standard of care (part 1) (Placebo Comparator): Placebo matching iptacopan standard of care
  Interventions: Drug: Placebo + standard of care
- Iptacopan + standard of care (part 2) (Active Comparator): Iptacopan + standard of care
  Interventions: Drug: Iptacopan (part 2)
- Iptacopan + placebo (part 2) (Active Comparator): Iptacopan + placebo standard of care
  Interventions: Drug: Iptacopan + placebo
- Placebo matching iptacopan + standard of care (part 2) (Active Comparator): Placebo matching iptacopan + standard of care
  Interventions: Drug: Placebo + standard of care

INTERVENTIONS:
Drug: Iptacopan (part 1) — Taken for 52 Weeks
  Other Names: LNP023
  Arms: Iptacopan + standard of care (part 1)
Drug: Iptacopan (part 2) — Taken for 52 Weeks
  Other Names: LNP023
  Arms: Iptacopan + standard of care (part 2)
Drug: Placebo + standard of care — Taken for 52 Weeks
  Arms: Placebo matching iptacopan + standard of care (part 1); Placebo matching iptacopan + standard of care (part 2)
Drug: Iptacopan + placebo — Taken for 52 Weeks
  Other Names: LNP023 and placebo
  Arms: Iptacopan + placebo (part 2)

SUMMARY:
The overall purpose of this two-part study is to evaluate the efficacy, safety and tolerability of iptacopan (LNP023) in addition to standard of care treatment.

DETAILED DESCRIPTION:
The overall purpose of this two-part study is to evaluate the efficacy, safety and tolerability of iptacopan (LNP023) in addition to standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

Unequivocally positive ANA test result and/or a positive anti dsDNA at screening Active biopsy-proven lupus nephritis within 3 months of screening demonstrating Class III or IV lupus nephritis with or without co-existing features of Class V lupus nephritis.

Documentation of active renal disease at the time of screening necessitating the commencement of therapy with corticosteroids in combination with MMF/MPS.

eGFR ≥ 30 ml/min/1.73 m2 Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infections Vaccination against Haemophilus influenzae infection Supportive care including stable dose regimen of anti-malarials (e.g. hydroxychloroquine) unless contraindicated, ACEi or ARB at either locally approved maximal daily dose or the maximally tolerated dose (per investigators' judgement) at screening, as per the local clinical practice. Doses should remain stable throughout the study.

First presentation or flare of lupus nephritis.

Exclusion Criteria:

Induction treatment with cyclophosphamide within 3 months of planned treatment for this study; treatment with calcineurin inhibitors within the previous 3 months prior to randomization.

Presence of rapidly progressive glomerulonephritis (RPGN) as defined by 50% decline in eGFR within 3 months prior to screening.

Renal biopsy presenting with interstitial fibrosis/tubular atrophy (IF/TA) or glomerulosclerosis of more than 50%, or which in the opinion of the investigator is such that it precludes likely response to immunosuppressive therapy.

Participants being treated with systemic corticosteroids (>5 mg/day prednisone or equivalent) for indications other than SLE or LN e.g. acute asthma, inflammatory bowel disease.

Participants being treated with systemic corticosteroids for SLE or LN will be excluded if they have taken more than an average of 15 mg/day prednisone (or equivalent) in the previous 4 weeks and more than an average of 30 mg/day in the previous 1 week Receipt of more than a total dose of 1000 mg equivalent i.v. pulse methylprednisolone (cumulative dose) within 2 weeks prior to enrollment (and at enrollment)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2028-09-28 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Proportion of patients achieving Complete Renal Response (CRR) at week 24 in the absence of renal flares | Baseline and week 24
  Part 1: To evaluate the proportion of patients achieving complete renal response with iptacopan treatment "A" plus standard of care, compared to treatment alone Part 2: To evaluate the proportion of patients achieving complete renal response with Iptacopan treatment "B" plus standard of care, compared to treatment "D" alone Part 2: To evaluate the proportion of patients achieving complete renal response with Iptacopan treatment "C" plus standard of care, compared to treatment "D" alone
  Complete Renal Response is defined as meeting the following criteria: estimated glomerular filtration rate (eGFR) ≥ 90 mL/min/1.73 m2 or no less than 85% of baseline value, and 24h urine protein-to-creatinine ratio (UPCR) ≤ 0.5 g/g.

SECONDARY OUTCOMES:
Parts 1 and 2: Proportion of patients achieving CRR or PRR in the absence of renal flares | Baseline, week 24, week 52
  Proportion of patients achieving complete renal response or partial renal response
Proportion of patients achieving ≥25% UPCR reduction in the absence of renal flares compared to baseline at week 24 | Baseline, week 24 week 52
  Frequency of renal flares between weeks 24 and 52
Log-transformed ratio to baseline of 24h UPCR at week 24 | Baseline week 24
  Dose exposure response for reduction in proteinurea. (each 24h urine protein-to-creatinine ratio value will based on two 24 urine collections sampled within 10 days before the respective study visit)
Change from baseline FACIT-Fatigue Score | Weeks 24 and 52
  Measure fatigue in patients
Change from baseline in SLEDAI-2K score at weeks 24 and 52 | Weeks 24 and 52
  Measure disease activity in SLE
Change from baseline in BILAG-2004 score at weeks 24 and 52 | Weeks 24 and 52
  Measure disease activity
Time-to-Complete Renal Response (CRR) based on first morning void(FMV) urine samples | Week 24 and Week 52
  Measurement of time to complete renal response based on urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (99):
- United States (25):
  - AKDHC Medical Research ServicesLLC, Phoenix, Arizona
  - Kaiser Permanente Fontana, Fontana, California
  - Univ Calif Irvine, Irvine, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Loma Linda University, San Bernardino, California
  - Olive View UCLA Medical Center, Sylmar, California
  - University of Colorado Denver, Aurora, Colorado
  - Royal Research Corp, Hollywood, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Nephrology Associates Of Central FL, Orlando, Florida
  - Florida Kidney Physicians, Riverview, Florida
  - Nep Assoc of Northern Illinois, Hinsdale, Illinois
  - Wichita Community Clcl Onco Program, Wichita, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Stony Brook Internists PC, East Setauket, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Dallas Nephrology Associates, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (3):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Brazil (6):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- China (6):
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shenzhen
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Montería
- France (4):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Ludwigshafen, Germany
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- India (7):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Puducherry
- Israel (3):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Malaysia (3):
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Taiping, Perak
  - Novartis Investigative Site, Selangor Darul Ehsan
- Mexico (4):
  - Novartis Investigative Site, Tampico, Tamaulipas
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Veracruz
- Philippines (3):
  - Novartis Investigative Site, Makati City, National Capital Region
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Quezon
- Portugal (5):
  - Novartis Investigative Site, Carnaxide
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- FDI Clinical Research, San Juan, Puerto Rico
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (5):
  - Novartis Investigative Site, Port de Sagunt, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Ciudad Real
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Bursa, Nilufer
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
- United Kingdom (2):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520